CLINICAL TRIAL: NCT04875026
Title: Frequency and Intensity of Local Reactions in Patients Treated With 4% 5-FU vs 4% 5-FU Associated With an Emollient Cream: a Randomised, Controlled Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: W00118 CR 401; 2020-000851-11 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-05-06 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This study is investigator-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 5-fluorouracil 4% (Tolak) + Dexeryl (Experimental): This group will apply 5-FU once daily for 4 weeks, and Dexeryl once daily for 8 weeks.
  Interventions: Drug: 5-fluorouracil 4% (Tolak); Device: Dexeryl
- 5-fluorouracil 4% (Tolak) (Other): This group will only apply 5-FU once daily for 4 weeks.
  Interventions: Drug: 5-fluorouracil 4% (Tolak)

INTERVENTIONS:
Drug: 5-fluorouracil 4% (Tolak) — Application of Tolak once daily in the evening for 4 weeks
Device: Dexeryl — Application of Dexeryl once daily in the morning for 8 weeks
  Arms: 5-fluorouracil 4% (Tolak) + Dexeryl

SUMMARY:
Transient local skin reactions with topical Actinic Keratosis treatments such as 5-FluoroUracil (5-FU) often lead to non-adhesion from patients and thus to treatment failure. In regards to 5-FU treatment, these local reactions are related to the pharmacological action of the molecule. The current therapeutic challenge is to reduce the local reactions induced by 5-FU without interfering with its efficacy, in particular by the use of an emollient cream.

The aim of the present study is to investigate how the use of an emollient, namely Dexeryl, could improve the local skin reactions occurring during 4 weeks of a 4% 5-FU treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible only if all of the following criteria apply:

Age

1. Participant must be more than 18 years old inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Individuals with a clinical diagnosis of actinic keratosis (AK).
3. Individuals harboring 5 or more clinically recognizable (palpable and/or visible to unaided eye) AK lesions of the face, and/or ears and/or scalp. The AK lesions must be clinically typical non hypertrophic and/or nonhyperkeratotic.
4. Subject in good general condition and free of any disease state or condition which, in the investigator's opinion, could impair evaluation of actinic keratosis or could expose the subject to an unacceptable risk by study participation.

   Sex
5. Male or female. A Female participant is eligible to participate if she is not a woman of childbearing potential (WOCBP), defined as postmenopausal (cessation of menses >12 months) or surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, total hysterectomy).

   Informed Consent
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Ethical/Legal considerations
7. Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. With AK lesions within treatment areas which are hyperkeratotic or which are clinically suspected to be squamous cell carcinoma (SCC).
2. With pre-existing local skin reactions with a total score ≥ 3.
3. History of hypersensitivity to the ingredients of Tolak® or Dexeryl®.
4. With a known allergy to peanut or soya.
5. Non postmenopausal or non surgically sterile woman considered as WOCBP, pregnant or breastfeeding women.

   Prior/Concomitant Therapy
6. Under systemic 5-fluorouracil or any systemic cancer treatment within eight weeks prior to the study.
7. Under any other topical AK treatments or therapies (e.g., Cryotherapy or Photodynamic therapy) in the treatment area(s) within eight weeks prior to starting the study.
8. Treated with systemic steroids, immunosuppressants or immunomodulators within four weeks prior to the study.
9. Under prescription retinoids or topical steroids in the treatment area(s) within four weeks prior to the study.
10. With known dihydropyrimidinedehydrogénase (DPD) deficiency or under treatment with brivudine, sorivudine or analogues within 4 weeks prior to starting the study.
11. Treated with glycolic acid products and alpha-hydroxy products in the treatment area(s) within four weeks prior to starting the study.
12. Treated with chemical peeling products in the treatment area(s) within eight weeks prior to starting the study.

    Prior/Concurrent Clinical Study Experience
13. Is participating in another clinical trial
14. Has participated in another clinical trial within the last 30 days, has received treatment with known remnant effects or undergone investigation liable to interfere with the present clinical trial Other Exclusions
15. Is a family member of the Investigator or any associate, colleague, and employee assisting in the conduct of the study (secretary, nurse, technician,…)
16. Is in a position likely to represent a conflict of interest
17. Has forfeited his / her freedom by administrative or legal award or is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Local Skin Reaction (LSR) total score | at 4 weeks or Last Observation Carried Forward (LOCF)
  Investigator-assessed score: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration) for a minimal score of 0 (best outcome possible), and a maximal score of 24 (worst outcome possible).

SECONDARY OUTCOMES:
Local Skin Reaction (LSR) total score | at 2 weeks (first follow-up)
  Investigator-assessed score: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration) for a minimal score of 0 (best outcome possible), and a maximal score of 24 (worst outcome possible).
Local Skin Reaction (LSR) total score | at 8 weeks (last follow up)
  Investigator-assessed score: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration) for a minimal score of 0 (best outcome possible), and a maximal score of 24 (worst outcome possible).
Local Skin Reaction (LSR) items alone | at 2 weeks (first follow-up)
  Presence/absence/intensity of each item of the LSR: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration). For each item, 0 is the best outcome possible, 4 is the worst
Local Skin Reaction (LSR) items alone | at 4 weeks (second follow up)
  Presence/absence/intensity of each item of the LSR: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration). For each item, 0 is the best outcome possible, 4 is the worst
Local Skin Reaction (LSR) items alone | at 8 weeks (last follow up)
  Presence/absence/intensity of each item of the LSR: 6 objective items scored from 0-4 (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration). For each item, 0 is the best outcome possible, 4 is the worst
Subjective signs at each visit | at 2 weeks (first follow-up)
  Patient questionnaire evaluating prurit (0-3), stinging/burning (0-3), pain (0-4). 0 is the best outcome, 10 is the worst outcome.
Subjective signs at each visit | at 4 weeks (second follow up)
  Patient questionnaire evaluating prurit (0-3), stinging/burning (0-3), pain (0-4). 0 is the best outcome, 10 is the worst outcome.
Subjective signs at each visit | at 8 weeks (last follow up)
  Patient questionnaire evaluating prurit (0-3), stinging/burning (0-3), pain (0-4). 0 is the best outcome, 10 is the worst outcome.
Local reactions according to Common Terminology Criteria for Adverse Event (CTCAE) grade 3 or 4 | at 2 weeks (first follow-up)
  Intensity grading of adverse events
Local reactions according to Common Terminology Criteria for Adverse Event (CTCAE) grade 3 or 4 | at 4 weeks (second follow up)
  Intensity grading of adverse events
Local reactions according to Common Terminology Criteria for Adverse Event (CTCAE) grade 3 or 4 | at 8 weeks (last follow up)
  Intensity grading of adverse events
Adverse Events reported by patients or noticed by investigator | at 2, 4 and 8 weeks (first follow-up)
Drop outs due to Adverse Events (AE) related to local skin reaction | at 2, 4 and 8 weeks (first follow-up)
  discontinuation rate
Use of rescue treatment | at 2 weeks (first follow-up)
Use of rescue treatment | at 4 weeks (second follow up)
Use of rescue treatment | at 8 weeks (last follow up)
Treatment satisfaction (acceptability): measured by Treatment Satisfaction Questionnaire for Medication version 9 (TSQM-9) | at 4 weeks (end of treatment) or at Patient Withdrawal
  The TSQM-9 questionnaire includes nine questions that assess patients' satisfaction by providing score on three scales: effectiveness (questions 1 to 3), convenience (questions 4 to 6) and global satisfaction (questions 7 to 9). The scores of each scale range from 0 to 100, where a higher score indicates a greater satisfaction
Treatment adherence | at 4 weeks
  assessed by the participant using a self questionnaire
Treatment adherence | at optional visit (when applicable), up to 8 weeks
  assessed by the participant using a self questionnaire
Health-related quality of life measured by actinic keratosis quality of life questionnaire (AKQoL) | at 8 weeks (last follow up)
  actinic keratosis quality of life patient questionnaire, for Spain and Germany only. 0 is the best outcome, 27 is the worst outcome
Rates of patients with complete and partial clearance rates | at 8 weeks (last follow up)
Rates of patients with partial clearance rates | at 8 weeks (last follow up)
Percentage change in number of AK lesions | at baseline
Percentage change in number of AK lesions | at 2 weeks (first follow-up)
Change in number of AK lesions | at 2 weeks (first follow-up)
Percentage change in number of AK lesions | at 4 weeks (second follow up)
Change in number of AK lesions | at 4 weeks (second follow up)
Percentage change in number of AK lesions | at 8 weeks (last follow up)
Change in number of AK lesions | at 8 weeks (last follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Eggert STOCKFLETH, Pr., Principal Investigator — Kath. Klinikum Bochum St. Josef-Hospital
Locations (27):
- France (5):
  - Private practice Maire, Arras
  - Chu de Nantes Hôtel-Dieu, Nantes
  - CHU Pau, Pau
  - CHU Poitiers, Poitiers
  - CHU St Etienne Hopital Nord, Saint-Etienne
- Germany (7):
  - Kath. Klinikum Bochum St. Josef-Hospital, Bochum
  - MVZ Dermatologisches Zentrum Bonn GmbH, Bonn
  - Private practice Quist, Bretzenheim
  - Private Practice Kurzen, Freising
  - Dermatologikum Hamburg, Hamburg
  - Hautarztpraxis, Witten
  - CentroDerm Clinic, Witten
- Italy (10):
  - Uni Clinic Brescia, Brescia
  - Uni Clinic Catania, Catania
  - Uni Clinic L'Aquila, Coppito
  - Policlinico San Martino, Genova
  - University of Messina, Messina
  - Uni Clinic Modena, Modena
  - NAPLES VANVITELLI UNIVERSITI (Federico II Hospital), Napoli
  - Azienda Unità Sanitaria Locale - IRCCS, Reggio Emilia
  - Catholic University Fondazione Policlinico Universitario A. Gemelli, Roma
  - Sapienza University of Rome - Polo Pontino, Terracina
- Spain (5):
  - Centre medic Congres, Barcelona
  - Hospital Alfredo Espinosa, Bilbao
  - Hospital Universitario Infanta Leonor, Madrid
  - Instituto Valenciano de Oncología,, Valencia
  - Hospital Marina Baixa, Villajoyosa

IPD SHARING:
Plan to Share IPD: No